CLINICAL TRIAL: NCT07334808
Title: Test-Retest Reliability of Grip Force Sense for Proprioception Assessment in Healthy Participants
Brief Title: Test-Retest Reliability of Grip Force Sense for Proprioception Assessment
Status: Recruiting | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Emrah Afsar, Assistant Professor, Kutahya Health Sciences University
Other Study IDs: 2025-a
Record Dates: First submitted 2025-12-31; First posted 2026-01-12 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Participants: Healthy volunteers. All participants will be assessed at baseline and re-assessed after a 1-week interval to determine test-retest reliability.

SUMMARY:
The aim of this study is to investigate the test-retest reliability of the grip force sense, a component of proprioception, using a dynamometer that is easily accessible and usable in a clinical setting. This provides an accessible assessment method for research in the field of proprioception.

DETAILED DESCRIPTION:
Participants aged 18-24 who are willing to participate in the study will be included. The necessary demographic information will be obtained using a data form. Participants will be seated in a chair with back support. Participants will perform isometric grip tasks with their arms at their sides, elbows flexed at 90°, and wrists in a neutral position. Subsequently, to assess participants' grip force sense, they will be measured on how accurately they can perform the applied 'force reproduction tasks'. Participants will be subjected to three different target force levels (10%, 30%, and 50% MVIC). A total of 9 trials will be conducted, with three repetitions for each force level. Participants will perform these 9 trials in two separate sessions (Session 1 and Session 2). The sessions will be conducted 7 days apart, in the same laboratory environment and by the same researcher. This will allow for the assessment of the test-retest reliability of the grip force sense. Throughout this process, grip strength will be measured using a digital hand dynamometer. Force values will be observed via a digital monitor. Three different error types will be calculated from the data related to the force reproduction task: (1) AE (Absolute Error), (2) CE (Constant Error), and (3) VE (Variable Error). Minimum-maximum values, mean and standard deviation will be used in the evaluation of continuous data, while frequency distributions and percentages will be used for categorical data. The data of the study will be analysed using IBM SPSS Statistics version 21.1 (IBM Corp., Armonk, NY) statistical package programmes. In all analyses, p<0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-24 years
* Volunteering to participate

Exclusion Criteria:

* Having a history of hand surgery
* Having any active pathology or pain complaints in the hand

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population consisted of healthy volunteers aged between 18 and 24 years without any history of previous hand surgery or presence of active pathology/pain in the hand.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2026-01-13 (Actual); Primary Completion 2026-12-12 (Estimated); Study Completion 2026-12-19 (Estimated)

PRIMARY OUTCOMES:
Absolute Error (AE) | Baseline and 1 week
  Absolute Error (AE) represents the absolute difference between the target force and the reproduced force, without regard to direction. It reflects the overall accuracy of the force reproduction task.
Constant Error (CE) | Baseline and 1 week
  Constant Error (CE) represents the directional difference between the target force and the reproduced force. It indicates the participant's directional bias (overshooting or undershooting the target).
Variable Error (VE) | Baseline and 1 week
  Variable Error (VE) represents the variability or consistency of the participant's performance across trials, regardless of the target. It reflects the consistency of force reproduction.

CONTACTS AND LOCATIONS:
Overall Officials: Emrah Afsar, Phd, Principal Investigator — Kutahya Health Science University
Locations (1):
- Kutahya Health Science University, Kütahya, Turkey (Türkiye)